CLINICAL TRIAL: NCT03238690
Title: Sequential Left Ventricular Assist Device (LVAD) Unloading and Conditioning to Induce Sustained Cardiac Recovery
Brief Title: LVAD Conditioning for Cardiac Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: STAVROS G DRAKOS (Other)
Responsible Party: Sponsor-Investigator, STAVROS G DRAKOS, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00095106
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: LVAD; Cardiac Recovery
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Controlled Cardiac Reloading (Experimental): Heart failure patients with recent LVAD implantation after an optimum unloading phase, will undergo controlled cardiac reloading through LVAD speed adjustment reductions in a controlled reloading phase
  Interventions: Device: Controlled Cardiac Reloading through LVAD Speed Adjustment

INTERVENTIONS:
Device: Controlled Cardiac Reloading through LVAD Speed Adjustment — LVAD speed is reduced at a fixed rate according to the particular LVAD device model implanted. LVAD speed reduction adjustments will be performed at visits occurring every 2 - 3 weeks, up to a total of 8 visits. Reduction of LVAD speed will continue until the soonest of: minimum operating setting as recommended in the LVAD Operator's manual is reached; the minimum setting tolerated by the subject is reached; the subject completes 8 visits; or until the subject receives a heart transplant.

SUMMARY:
The purpose of this study is to investigate the potential recovery of heart function in end-stage heart failure patients supported with a Left Ventricular Assist Device (LVAD) through applying a myocardial conditioning protocol. During myocardial conditioning, LVAD speed is reduced gradually in order to increase the work load of the heart. Multiple previous studies have shown that interventions like this may improve heart function and give patients the opportunity for a better quality of life.

DETAILED DESCRIPTION:
Heart failure can be caused by various disorders, such as myocardial infarction, hypertension, viral infection, exposure to toxins, chemotherapy, or genetically transmitted muscular diseases. Regardless of the etiology, these disorders initiate ventricular remodeling, an adaptive, compensatory process which becomes progressively maladaptive and the cause of functional and clinical deterioration, eventually leading to heart failure. Local and systemic compensatory responses that initially allow surviving muscle to maintain hemodynamic function continue over time and due to this persistent compensatory over-activity the initially unaffected myocardium becomes dysfunctional. These compensatory responses to an abnormal cardiac load or myocardial injury involve several pathophysiological adaptations in the cardiac structure at the genetic, molecular, cellular, and tissue levels. Furthermore, left ventricular pressure and volume overload has shown to alter metabolic substrate utilization, decrease mitochondrial function and reduce energy production in the failing heart.

Mechanical circulatory support with LVAD has become a standard bridge to cardiac transplantation, and has also been approved in the United States as permanent (destination) therapy for selected patients presenting with end-stage heart failure. Clinical experience with LVAD support has shown that it can reverse the complex process of chronic left ventricular remodeling to a point where a subset of patients could be weaned from the device after restoration of basic cardiac function. LVAD-induced mechanical unloading of the failing heart leads to reduced mitochondrial density, structure and function, and interventions that enhance mitochondrial biogenesis, function and structure, such as controlled cardiac reloading may enhance LVAD-induced myocardial reverse remodeling and cardiac recovery. This study is designed to investigate gradual reduction in LVAD speed within the range defined by the assist device manufacturer's manual as appropriate for regular clinic use, to determine the effect on reverse remodeling and myocardial recovery in end-stage heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure undergoing LVAD implantation as a bridge to transplant
* Enrolled in the Effects of Mechanical Unloading on Myocardial Function and Structure study (IRB 30622)

Exclusion Criteria:

* Neither the subject nor the subject's representative is willing to provide written consent for participation
* Subjects with adverse events leading to hospitalization during the optimum unloading phase are excluded from participation in the controlled reloading phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline (prior to LVAD implantation) and 12 months post-LVAD implantation, or at time of LVAD explantation/heart transplant
  LVEF is measured by echocardiography. The average change in LVEF from baseline to 12 months or transplant in the study participant arm will be compared to results from an historical control group.

SECONDARY OUTCOMES:
Change in Left Ventricular End Diastolic Diameter (LVEDD) | Baseline (prior to LVAD implantation) and 12 months post-LVAD implantation, or at time of LVAD explantation/heart transplant
  LVEDD is measured by echocardiography. The average change in LVEDD from baseline to 12 months or transplant in the study participant arm will be compared to results from an historical control group.
Change in Left Ventricular End Systolic Diameter (LVESD) | Baseline (prior to LVAD implantation) and 12 months post-LVAD implantation, or at time of LVAD explantation/heart transplant
  LVESD is measured by echocardiography. The average change in LVESD from baseline to 12 months or transplant in the study participant arm will be compared to results from an historical control group.
Change in Left Ventricular End Diastolic Volume (LVEDV) | Baseline (prior to LVAD implantation) and 12 months post-LVAD implantation, or at time of LVAD explantation/heart transplant
  LVEDV is measured by echocardiography. The average change in LVEDV from baseline to 12 months or transplant in the study participant arm will be compared to results from an historical control group.
Change in Left Ventricular End Systolic Volume (LVESV) | Baseline (prior to LVAD implantation) and 12 months post-LVAD implantation, or at time of LVAD explantation/heart transplant
  LVESV is measured by echocardiography. The average change in LVESV from baseline to 12 months or transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose 1-phosphate levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for Glucose 1-phosphate levels. The average change in Glucose 1-phosphate from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose 6-phosphate levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for Glucose 6-phosphate levels. The average change in Glucose 6-phosphate from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Pyruvate levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for Pyruvate levels. The average change in Pyruvate from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Lactic Acid levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for Lactic Acid levels. The average change in Lactic Acid from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Acetyl Coenzyme A levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for Acetyl Coenzyme A levels. The average change in Acetyl Coenzyme A from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose Transporter 1 (GLUT1) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for GLUT1 levels. The average change in GLUT1 from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose Transporter 1 (GLUT1) messenger ribonucleic acid (mRNA) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for GLUT1 mRNA levels. The average change in GLUT1 mRNA from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose Transporter 4 (GLUT4) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for GLUT4 levels. The average change in GLUT4 from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Glucose Transporter 4 (GLUT4) messenger ribonucleic acid (mRNA) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for GLUT4 mRNA levels. The average change in GLUT4 mRNA from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Mitochondrial Pyruvate Carrier 1 (MPC1) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for MPC1 levels. The average change in MPC1 from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Mitochondrial Pyruvate Carrier 2 (MPC2) levels | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for MPC2 levels. The average change in MPC2 from baseline to transplant in the study participant arm will be compared to results from an historical control group.
Change in heart tissue Mitochondrial Density | Baseline (LVAD implantation) and at time of LVAD explantation/heart transplantation (up to 12 months)
  Heart tissue samples will be collected at LVAD implantation when the tissue from the core becomes available and then at explant when the whole heart becomes available, and will be analyzed for mitochondrial density by electron microscopy. The average change in mitochondrial density from baseline to transplant in the study participant arm will be compared to results from an historical control group.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Drakos, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George RS, Sabharwal NK, Webb C, Yacoub MH, Bowles CT, Hedger M, Khaghani A, Birks EJ. Echocardiographic assessment of flow across continuous-flow ventricular assist devices at low speeds. J Heart Lung Transplant. 2010 Nov;29(11):1245-52. doi: 10.1016/j.healun.2010.05.032. Epub 2010 Aug 5. PMID 20688540
- [Background] Healy AH, Koliopoulou A, Drakos SG, McKellar SH, Stehlik J, Selzman CH. Patient-controlled conditioning for left ventricular assist device-induced myocardial recovery. Ann Thorac Surg. 2015 May;99(5):1794-6. doi: 10.1016/j.athoracsur.2014.07.058. PMID 25952209
- [Background] Frazier OH, Baldwin AC, Demirozu ZT, Segura AM, Hernandez R, Taegtmeyer H, Mallidi H, Cohn WE. Ventricular reconditioning and pump explantation in patients supported by continuous-flow left ventricular assist devices. J Heart Lung Transplant. 2015 Jun;34(6):766-72. doi: 10.1016/j.healun.2014.09.015. Epub 2014 Sep 28. PMID 25447571